CLINICAL TRIAL: NCT00389168
Title: Randomized, Double-blind Evaluation of the Effects of Irbesartan and Atenolol on Cardiovascular Structure and Function in Subjects With Hypertension and Left Ventricular Hypertrophy
Brief Title: Irbesartan and Atenolol in Hypertensive Heart Disease
Acronym: SILVHIA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Bristol-Myers Squibb (Industry); Sanofi (Industry); Swedish Heart Lung Foundation (Other)
Responsible Party: Principal Investigator, Thomas Kahan, Professor, Principal investigator and Study Chair, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV131-052
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Results first posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Hypertension
Keywords: Hypertension; Cardiac hypertrophy; Angiotensin; Human
MeSH Terms: conditions — Hypertension; Cardiomegaly | interventions — Irbesartan; Atenolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Irbesartan (Experimental): Irbesartan per os titrated to 300 mg od, 48 weeks
  Interventions: Drug: Irbesartan
- Atenolol (Active Comparator): Atenolol per os titrated to 100 mg od, 48 weeks
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Irbesartan — Titrated to 300 mg od, 48 weeks.
  Other Names: Aprovel
  Arms: Irbesartan
Drug: Atenolol — Titrated to 100 mg od, 48 weeks.
  Other Names: Tenormin
  Arms: Atenolol

SUMMARY:
The renin-angiotensin-aldosterone system has been implicated in the control of structural changes of the heart and the vasculature, beyond the effects on blood pressure.

This projects examines the importance of the renin-angiotensin-aldosterone system and the sympathetic nervous system in the control of cardiac and vascular structure and function in subjects with hypertension.Patients with hypertension and left ventricular hypertrophy were randomized to an angiotensin receptor blocker or a beta adrenergic receptor blocker for 48 weeks. Repeat investigations of blood pressure, structure and function of the heart and the vascular tree, and neurohormones were performed. Two control groups, consisting of normotensive subjects and of hypertensive subjects with no cardiac hypertrophy were also examined for comparison.

DETAILED DESCRIPTION:
We included 115 patients with hypertension and cardiac hypertrophy, established by echocardiography. Extensive echocardiographic examinations, ultrasonography of the carotid arteries, 24h Holter registrations, 24h ambulatory blood pressure monitoring monitoring, neurohormones and blood samples for inflammation and hemostasis markers and endothelial function were done at weeks 0, 12, 24, and 48. Matched control groups (1:3, i.e. 38 normotensive subjects and 38 hypertensive subjects with no signs of hypertensive heart disease were examined at one occasion. All patients obtained irbesartan or atenolol for 12 weeks; a diuretic and a calcium antagonist was added when needed thereafter in order to obtained a blood pressure below 140/90 mm Hg. All analyses were performed central in a core laboratory.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 ys old
* Male or female with no child bearing potential
* Seated blood pressure diastolic 90-115 mm Hg
* Left ventricular mass above 131 g/m2 for men, above 100 g/m2 for women
* Informed consent

Exclusion Criteria:

* Coronary artery disease, heart failure or other significant cardiac disorder
* Cerebrovascular accident within the past 6 months
* A seated systolic blood pressure above 200 mm Hg
* Significant renal disease, collagen or vascular disease, or gastrointestinal condition
* Significant allergy or intolerance to study drug
* Alcohol or drug abuse
* Uncontrolled diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 1995-04; Primary Completion 1997-04 (Actual); Study Completion 1997-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kahan, MD, PhD, Study Chair — Karolinska Institutet, Department of Clinical Sciences, Danderyd Hospital, SE-182 88 Stockholm, Sweden
Locations (1):
- Karolinska Institutet, Daprtment of Clinical Sciences, Danderyd Hospital, Cardiovascular Research Laboratory, Stockholm, Sweden

REFERENCES:
- [Result] Malmqvist K, Kahan T, Edner M, Held C, Hagg A, Lind L, Muller-Brunotte R, Nystrom F, Ohman KP, Osbakken MD, Ostergern J. Regression of left ventricular hypertrophy in human hypertension with irbesartan. J Hypertens. 2001 Jun;19(6):1167-76. doi: 10.1097/00004872-200106000-00023. PMID 11403367
- [Result] Nystrom F, Malmqvist K, Ohman KP, Kahan T. Nurse-recorded and ambulatory blood pressure predicts treatment-induced reduction of left ventricular hypertrophy equally well in hypertension: results from the Swedish irbesartan left ventricular hypertrophy investigation versus atenolol (SILVHIA) study. J Hypertens. 2002 Aug;20(8):1527-33. doi: 10.1097/00004872-200208000-00015. PMID 12172314
- [Result] Malmqvist K, Kahan T, Edner M, Bergfeldt L. Comparison of actions of irbesartan versus atenolol on cardiac repolarization in hypertensive left ventricular hypertrophy: results from the Swedish Irbesartan Left Ventricular Hypertrophy Investigation Versus Atenolol (SILVHIA). Am J Cardiol. 2002 Nov 15;90(10):1107-12. doi: 10.1016/s0002-9149(02)02777-7. PMID 12423712
- [Result] Malmqvist K, Ohman KP, Lind L, Nystrom F, Kahan T. Long-term effects of irbesartan and atenolol on the renin-angiotensin-aldosterone system in human primary hypertension: the Swedish Irbesartan Left Ventricular Hypertrophy Investigation versus Atenolol (SILVHIA). J Cardiovasc Pharmacol. 2003 Dec;42(6):719-26. doi: 10.1097/00005344-200312000-00005. PMID 14639093
- [Result] Muller-Brunotte R, Kahan T, Malmqvist K, Ring M, Edner M. Tissue velocity echocardiography shows early improvement in diastolic function with irbesartan and atenolol therapy in patients with hypertensive left ventricular hypertrophy. Results form the Swedish Irbesartan Left Ventricular Hypertrophy Investigation vs Atenolol (SILVHIA). Am J Hypertens. 2006 Sep;19(9):927-36. doi: 10.1016/j.amjhyper.2006.02.009. PMID 16942935
- [Result] Mortsell D, Malmqvist K, Held C, Kahan T. Irbesartan reduces common carotid artery intima-media thickness in hypertensive patients when compared with atenolol: the Swedish Irbesartan Left Ventricular Hypertrophy Investigation versus Atenolol (SILVHIA) study. J Intern Med. 2007 May;261(5):472-9. doi: 10.1111/j.1365-2796.2007.01775.x. PMID 17444886
- [Result] Malmqvist K, Kahan T, Edner M, Bergfeldt L. Cardiac repolarization and its relation to ventricular geometry and rate in reverse remodelling during antihypertensive therapy with irbesartan or atenolol: results from the SILVHIA study. J Hum Hypertens. 2007 Dec;21(12):956-65. doi: 10.1038/sj.jhh.1002250. Epub 2007 Jul 19. PMID 17637792
- [Result] Muller-Brunotte R, Kahan T, Lopez B, Edner M, Gonzalez A, Diez J, Malmqvist K. Myocardial fibrosis and diastolic dysfunction in patients with hypertension: results from the Swedish Irbesartan Left Ventricular Hypertrophy Investigation versus Atenolol (SILVHIA). J Hypertens. 2007 Sep;25(9):1958-66. doi: 10.1097/HJH.0b013e3282170ada. PMID 17762662
- [Result] Kurland L, Hallberg P, Melhus H, Liljedahl U, Hashemi N, Syvanen AC, Lind L, Kahan T. The relationship between the plasma concentration of irbesartan and the antihypertensive response is disclosed by an angiotensin II type 1 receptor polymorphism: results from the Swedish Irbesartan Left Ventricular Hypertrophy Investigation vs. Atenolol (SILVHIA) Trial. Am J Hypertens. 2008 Jul;21(7):836-9. doi: 10.1038/ajh.2008.190. Epub 2008 May 8. PMID 18464745
- [Result] Liljedahl S, Kahan T, Lind L, Arnlov J. The effects of antihypertensive treatment on the doppler-derived myocardial performance index in patients with hypertensive left ventricular hypertrophy: results from the Swedish irbesartan in left ventricular hypertrophy investigation versus atenolol (SILVHIA). Echocardiography. 2009 Aug;26(7):753-8. doi: 10.1111/j.1540-8175.2008.00886.x. PMID 19486119
- [Result] Muller-Brunotte R, Kahan T, Malmqvist K, Edner M; Swedish ibesartan left ventricular hypertrophy investigation vs atenolol (SILVHIA). Blood pressure and left ventricular geometric pattern determine diastolic function in hypertensive myocardial hypertrophy. J Hum Hypertens. 2003 Dec;17(12):841-9. doi: 10.1038/sj.jhh.1001622. PMID 14704728
- [Result] Muller-Brunotte R, Edner M, Malmqvist K, Kahan T. Irbesartan and atenolol improve diastolic function in patients with hypertensive left ventricular hypertrophy. J Hypertens. 2005 Mar;23(3):633-40. doi: 10.1097/01.hjh.0000160222.17092.b8. PMID 15716707
- [Result] Jekell A, Malmqvist K, Wallen NH, Mortsell D, Kahan T. Markers of inflammation, endothelial activation, and arterial stiffness in hypertensive heart disease and the effects of treatment: results from the SILVHIA study. J Cardiovasc Pharmacol. 2013 Dec;62(6):559-66. doi: 10.1097/FJC.0000000000000017. PMID 24084214
- [Result] Kurland L, Liljedahl U, Karlsson J, Kahan T, Malmqvist K, Melhus H, Syvanen AC, Lind L. Angiotensinogen gene polymorphisms: relationship to blood pressure response to antihypertensive treatment. Results from the Swedish Irbesartan Left Ventricular Hypertrophy Investigation vs Atenolol (SILVHIA) trial. Am J Hypertens. 2004 Jan;17(1):8-13. doi: 10.1016/j.amjhyper.2003.09.009. PMID 14700505

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter Swedish study. Patients with primary hypertension and left ventricular (LV) hypertrophy.
Pre-assignment Details: All participants received a placebo washout period during 4 weeks at the beginning of the study.
  One patient of the 115 included was during the course of the study diagnosed with Mb Conn (adrenal tumor causing endocrine secondary hypertension). This patient was excluded from all analyses. Thus, there are 114 patients included in the dataset.
Groups:
- Irbesartan; Atenolol: A double blind study with parallel group treatment with irbesartan or atenolol; addition of hydrochlorothiazide (HCTZ) and felodipine when needed to achieve < 140/90 mm Hg
Period: Overall Study
Arm/Group | Irbesartan | Atenolol
Started | 56 | 58
Completed | 47 | 53
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Atenolol; Irbesartan: A double blind study with parallel group treatment with irbesartan or atenolol; addition of HCTZ and felodipine when needed to achieve < 140/90 mm Hg
- Total: Total of all reporting groups
Arm/Group | Atenolol | Irbesartan | Total
Number analyzed (Participants) | 58 | 56 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 49 | 100
  >=65 years | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10) | 54 (8) | 54 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 40 | 36 | 76
Region of Enrollment [Number; unit: participants]
  Sweden | 58 | 56 | 114

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Safety was assessed by non-directed questions, and all observed and volunteered adverse events were recorded at each study visit. Serious adverse events were defined by, and reported according to the regulations of good clinical practice (GCP). none were considered related to the study medication.
Time Frame: Treatment period was baseline to 48 weeks
Measure: Number; unit: Participants
Arm/Group | Atenolol | Irbesartan
Number analyzed (Participants) | 58 | 56
Participants | 5 | 5

2. Primary Outcome: Changes in Left Ventricular Mass Index
Description: Repeated measures multivariate analysis of variance (MANOVA) at time points 0, 12, 24, and 48 weeks. Data are presented as left ventricular mass in gram (g) indexed for body mass index (in m^2).
Time Frame: Baseline and 48 weeks
Population: Data on echocardiography is not always available at all time points and for all participants. This is reflected by the number of observations, which sometimes are less than the number of participants.
Measure: Mean (95% Confidence Interval); unit: g/m^2
Arm/Group | Atenolol | Irbesartan
Number analyzed (Participants) | 50 | 44
g/m^2
  12 weeks | -1 [-6 to 4] | -9 [-15 to -6]
  24 weeks | -6 [-12 to 0] | -14 [-22 to -6]
  48 weeks | -14 [-20 to 9] | -26 [-34 to -18]

3. Secondary Outcome: Left Ventricular Diastolic Function Assessed by the E/A Ratio
Description: Changes in left ventricular diastolic function from baseline to week 48 will be evaluated as the difference in E/A ratio. Conventional pulsed wave Doppler echocardiography was used for recordings of mitral inflow in. The peak of early (E) and late (A) mitral flow velocities were measured, and the E/A-ratio was calculated. Repeated measures MANOVA at time points 0, 12, 24, and 48 weeks. Some echocardiographic recordings at some time point may be of insufficient quality or missing, and the number of observations may not always correspond to the total number of participants at all time points.
Time Frame: Baseline to 48 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Atenolol | Irbesartan
Number analyzed (Participants) | 50 | 45
ratio
  Week 12 | 0.18 (0.23) | 0.10 (0.22)
  Week 24 | 0.16 (0.28) | 0.04 (0.18)
  Week 48 | 0.13 (0.24) | 0.10 (0.21)

4. Secondary Outcome: Blood Pressure
Description: Difference in Diastolic Blood Pressure. Repeated measures multivariable analysis of variance (MANOVA) at time points 0, 12, 24, and 48 weeks
Time Frame: Baseline to 48 weeks
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Atenolol | Irbesartan
Number analyzed (Participants) | 53 | 47
mm Hg | -16.3 [-18.5 to -14.0] | -18.8 [-21.4 to -16.3]

5. Secondary Outcome: Changes of Venous Plasma Angiotensin II as a Marker of the Renin-Angiotensin-Aldosterone System
Description: Venous plasma concentrations of angiotensin II were measured in order to study the possible associations between the activity of the renin-angiotensin-aldosteone system and changes in left ventricular mass. Further analyses of other components of the renin-angiotensin-aldosterone system and of other hormonal system (e.g. the sympathetic nervous system) have also been performed and published. Repeated measures MANOVA at time points 0, 12, 24, and 48 weeks. Data were log-transformed to avoid skewness before statistical evaluation. However, tabular data are given as mean values with 95% confidence to improve readability.
Time Frame: Baseline to 48 weeks
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Atenolol | Irbesartan
Number analyzed (Participants) | 53 | 46
pmol/L
  Weel 12 | -1.0 [-1.4 to -0.5] | 3.0 [1.2 to 4.9]
  Week 24 | -0.8 [-1.4 to -0.1] | 3.3 [1.8 to 4.7]
  Week 48 | -0.2 [-0.9 to 0.4] | 10.0 [5.0 to 15.0]

6. Secondary Outcome: Effects on Carotid Artery Wall Thickness
Description: Changes in common carotid artery intima-media thickness, assessed by ultrasonography.
Time Frame: Baseline to 48 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Atenolol | Irbesartan
Number analyzed (Participants) | 56 | 52
mm | 0.03 (0.12) | -0.01 (0.10)

ADVERSE EVENTS:
Time Frame: The entire duration of study: that is 4-6 weeks of single-blinded placebo run-in, 48 weeks of double-blinded medication, and 4 weeks following completion of the study.
Description: Defied and reported according to study protocol.
Groups:
- Irbesratan; Atenolol: A double blind study with parallel group treatment with irbesartan or atenolol; addition of HCTZ and felodipine when needed to achieve < 140/90 mm Hg
Arm/Group | Irbesratan | Atenolol
Serious Adverse Events (participants affected / at risk) | 5/56 | 5/58
Other Adverse Events (participants affected / at risk) | 0/56 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irbesratan (N=56) | Atenolol (N=58)
inadequate blood pressure reduction (Cardiac disorders) | 2 (2) | 0 (0) — None of withdrawals were considered likely related to the drugs studied.
events were not documented specifically in the records available (Social circumstances) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less